CLINICAL TRIAL: NCT00368238
Title: Effects of Recombinant Human Erythropoietin on Platelet Function in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Heart Association (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0506000139; AHA 0555844T
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2006-08-24 (Estimated); Status verified 2006-08

CONDITIONS: Healthy Subjects
Keywords: Platelet function tests; Erythropoietin; Aspirin; Clopidogrel
MeSH Terms: interventions — Pharmaceutical Preparations; Aspirin; Clopidogrel

INTERVENTIONS:
Drug: Recombinant human erythropoietin alfa (drug)
Drug: Aspirin (drug)
Drug: Clopidogrel (drug)

SUMMARY:
The purpose of this study is to see if a naturally-occurring hormone called erythropoietin changes the action of platelets in the blood. Erythropoietin is made by the kidneys to stimulate red blood cell production to prevent anemia. Platelets are small cells in the blood that help clot blood in case of injury. Platelets also sometimes form blood clots in blood vessels that may cause heart attacks. This study is trying to determine whether erythropoietin increases the clotting action of platelets. Information on erythropoietin in healthy subjects may eventually help in the treatment of patients with heart attacks.

DETAILED DESCRIPTION:
Anti-apoptotic effects of erythropoietin in experimental myocardial infarction and ischemia-reperfusion injury suggest potential for therapeutic benefit in patients with acute MI. Before the therapeutic potential of rHuEpo in acute MI can be tested in large clinical trials, more information on the effects of short-term rHuEpo on platelet function are needed. Accordingly, the current proposal aims to determine the effects of 3 doses of rHuEpo (100U/kg, 200U/kg and 400U/kg daily for 3 days) on platelet function and other safety measures in healthy subjects.

Specific Aim: To determine the effects of three ascending doses of rHuEpo vs. placebo on in vivo and in vitro platelet function in healthy subjects treated with aspirin and clopidogrel.

Hypotheses to be tested: 1) 1) Short-term administration of rHuEpo does not alter bleeding time responses to aspirin and clopidogrel when compared with placebo. 2) Short-term administration does not alter in vitro platelet aggregation responses to aspirin and clopidogrel when compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-40 years
* Able and willing to provide written informed consent
* Bleeding time <10 minutes

Exclusion Criteria:

* Any chronic medical disease
* Chronic or frequent over-the-counter or prescription medication use
* Hemoglobin >15 gm/dl for both genders or <13 gm/dl (men) or <12 gm/dl (women)
* Platelet count >400,000/µl or <150,000/µl
* Blood pressure > 140/90 mmHg

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96
Dates: Start 2005-10; Study Completion 2006-07

PRIMARY OUTCOMES:
Bleeding time
Platelet function assay closure time

SECONDARY OUTCOMES:
Complete Blood Count
PT
PTT
P-selectin
von Willebrand factor

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Katz, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States